CLINICAL TRIAL: NCT00439647
Title: A Two Year Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Fracture Efficacy and Safety of Intravenous Zoledronic Acid 5 mg Annually for the Treatment of Osteoporosis in Men
Brief Title: Efficacy in Reducing Fractures and Safety of Zoledronic Acid in Men With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446M2309
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2011-11-16 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2011-10

CONDITIONS: Male Osteoporosis
Keywords: Osteoporosis; males; vertebral fractures; clinical fractures; bone mineral density; bone biomarkers; zoledronic acid
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic Acid (Experimental): 5 mg/100 ml administered via a peripheral intravenous site as a slow infusion over 15 minutes. The intravenous (i.v.) infusion was delivered via vented infusion line (to allow constant flow) and 20-22 gauge angiocatheter, and preceded and followed by a 10 ml normal saline flush of the intravenous line for a total volume infused of 120 ml once a year.
  Interventions: Drug: Zoledronic acid 5 mg iv
- Placebo (Placebo Comparator): 100 ml Placebo administered via a peripheral intravenous site as a slow infusion over 15 minutes. The i.v. infusion was delivered via vented infusion line (to allow constant flow) and 20-22 gauge angiocatheter, and preceded and followed by a 10 ml normal saline flush of the intravenous line for a total volume infused of 120 ml once a year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid 5 mg iv — Zoledronic acid 5 mg iv given once a year.
  Other Names: Aclasta,; Reclast
  Arms: Zoledronic Acid
Drug: Placebo — Placebo intravenous (i.v.) once a year
  Arms: Placebo

SUMMARY:
This study will investigate if the drug zoledronic acid given once yearly is safe and has beneficial effects in treating osteoporosis by reducing bone loss and fractures in men with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

• Osteoporosis as defined by very low bone mineral density in the hip and spine or low bone mineral density in the hip combined with presence of 1-3 mild or moderate fractures of the vertebrae

Exclusion Criteria:

* Low Vitamin D
* Renal insufficiency
* Previous treatment with certain anti-osteoporotic therapies (except after certain washout periods): calcitonin, bisphosphonates, parathyroid hormone (PTH), sodium fluoride, strontium ranelate,
* Previous treatment with testosterone, anabolic steroids or growth hormone
* Chronic use of systemic corticosteroids (oral or i.v.) within the last year
* History of any cancer or metastases within the last 5 years
* History of brittle bone disease, multiple myeloma, or Paget's disease, or any other metabolic bone disease, except osteoporosis
* Bilateral hip replacements

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1199 (Actual)
Dates: Start 2006-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Argentina; Novartis Pharmaceuticals, Principal Investigator — Novartis Belgium; Novartis Pharmaceuticals, Principal Investigator — Novartis Brazil; Novartis Pharmaceuticals, Principal Investigator — Novartis Czech Republic; Novartis Pharmaceuticals, Principal Investigator — Novartis Denmark; Novartis Pharmaceuticals, Principal Investigator — Novartis Finland; Novartis Pharmaceuticals, Principal Investigator — Novartis Germany; Novartis Pharmaceuticals, Principal Investigator — Novartis Hungary; Novartis Pharmaceuticals, Principal Investigator — Novartis Norway; Novartis Pharmaceuticals, Principal Investigator — Novartis Portugal; Novartis Pharmaceuticals, Principal Investigator — Novartis Romania; Novartis Pharmaceuticals, Principal Investigator — Novartis Spain; Novartis Pharmaceuticals, Principal Investigator — Novartis Slovakia; Novartis Pharmaceuticals, Principal Investigator — Novartis Sweden; Novartis Pharmaceuticals, Principal Investigator — Novartis; Novartis Pharmaceuticals, Principal Investigator — Novartis United Kingdom; Novartis Pharmaceuticals, Principal Investigator — Novartis Australia; Novartis Pharmaceuticals, Principal Investigator — Novartis Italy; Novartis Pharmaceuticals, Principal Investigator — Novartis Austria; Novartis Pharmaceuticals, Principal Investigator — Novartis Iceland; Novartis Pharmaceuticals, Principal Investigator — Novartis Poland; Novartis Pharmaceuticals, Principal Investigator — Novartis Russia; Novartis Pharmaceuticals, Principal Investigator — Novartis (South Africa)
Locations (128):
- Argentina (4):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mar del Plata
  - Novartis Investigative Site, San Miguel de Tucumán
- Australia (3):
  - Novartis Investigative Site, Geelong-VIC
  - Novartis Investigative Site, Maroochydore-QLD
  - Novartis Investigative Site, Randwick-NSW
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (11):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Diepenbeek
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, Gozée
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Merksem
  - Novartis Investigative Site, Wilrijk
- Brazil (4):
  - Novartis Investigative Site, Brasília
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Czechia (4):
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- Denmark (5):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Odense C
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- Germany (16):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Bad Pyrmont
  - Novartis Investigative Site, Braunfels
  - Novartis Investigative site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kempen
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Veszprém
- Novartis Investigative site, Kopavogur, Iceland
- Italy (3):
  - Novartis Investigative site, Arenzano
  - Novartis Investigative site, Siena-SI
  - Novartis Investigative site, Valeggio sul Mincio
- Norway (6):
  - Novartis Investigative Site, Elverum
  - Novartis Investigative Site, Gjettum
  - Novartis Investigative Site, Hamar
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Paradis
  - Novartis Investigative Site, Trondheim
- Poland (2):
  - Novartis Investigative site, Bialystok
  - Novartis Investigative site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Russia (5):
  - Novartis Investigative site, Moscow
  - Novartis Investigative site, Saint Petersburg
  - Novartis Investigative site, Tyumen
  - Novartis Investigative site, Yaroslavl
  - Novartis Investigative site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative site, Ľubochňa
  - Novartis Investigative Site, Piešťany
- South Africa (3):
  - Novartis Investigative site, Cape Town
  - Novartis Investigative site, Rosebank-Johannesburg
  - Novartis Investigative site, Western Cape
- Spain (15):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, L'Hospitalet de Llobregat
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Mérida
  - Novartis Investigative Site, Oviedo
  - Novartis Investigative Site, Sabadell
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Villajoyosa
- Sweden (8):
  - Novartis investigative site, Gothenburg
  - Novartis investigative site, Linköping
  - Novartis investigative site, Lund
  - Novartis investigative site, Malmo
  - Novartis investigative site, Örebro
  - Novartis investigative site, Stockholm
  - Novartis investigative site, Umeå
  - Novartis investigative site, Uppsala
- Switzerland (8):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Baden
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative site, Sion
  - Novartis Investigative Site, Zurich
- United Kingdom (11):
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative site, Chorley
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middx
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Penarth
  - Novartis Investigative site, Reading-Berkshire

REFERENCES:
- [Derived] Boonen S, Reginster JY, Kaufman JM, Lippuner K, Zanchetta J, Langdahl B, Rizzoli R, Lipschitz S, Dimai HP, Witvrouw R, Eriksen E, Brixen K, Russo L, Claessens F, Papanastasiou P, Antunez O, Su G, Bucci-Rechtweg C, Hruska J, Incera E, Vanderschueren D, Orwoll E. Fracture risk and zoledronic acid therapy in men with osteoporosis. N Engl J Med. 2012 Nov 1;367(18):1714-23. doi: 10.1056/NEJMoa1204061. PMID 23113482

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 100 ml Placebo administered via a peripheral intravenous site as a slow infusion over 15 minutes. The intravenous (i.v.) infusion was delivered via vented infusion line (to allow constant flow) and 20-22 gauge angiocatheter, and preceded and followed by a 10 ml normal saline flush of the intravenous line for a total volume infused of 120 ml once a year.
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 588 ("Started" indicates intent to treat (ITT) and safety set.) | 611
Modified Intent to Treat (mITT) | 553 | 574
Completed | 530 | 540
Not Completed | 58 | 71
Not completed — Withdrawal by Subject | 25 | 22
Not completed — Death | 15 | 18
Not completed — Adverse Event | 11 | 11
Not completed — Lost to Follow-up | 4 | 12
Not completed — Protocol Violation | 3 | 4
Not completed — Lack of Efficacy | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 588 | 611 | 1199
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.3) | 65.7 (8.6) | 65.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 588 | 611 | 1199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One New Morphometric Vertebral Fracture Over 24 Months
Description: Vertebral fracture (VF) was assessed based on morphometry. QM(quantitative morphometry) incident VF(QM positive) is defined by at least 20% decrease in vertebral height of at least 4mm. If participant had QM positive at any vertebrae at any visit, x-rays from visits for participants were evaluated using Genant semi-quantitative method for VF assessment: Grade1 Mild VF is defined as 20-24% decrease in anterior, middle, and/or posterior vertebral height. Grade2 moderate VF is defined as 25-40% decrease in vertebral height. Grade3 Severe VF is defined as more than 40% decrease in vertebral height
Time Frame: 24 Months
Population: Modified Intent-to-treat (mITT) population included all randomized subjects who had a baseline and at least one post-baseline assessment of the primary efficacy variable. In this analysis, missing Month 24 fractures were imputed using LOCF.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of Participants | 1.6 | 4.9

2. Secondary Outcome: Percentage of Participants With at Least One New Morphometric Vertebral Fracture Over 12 Months
Description: as for outcome 1
Time Frame: 12 Months
Population: Modified Intent-to-treat (mITT) population included all randomized subjects who had a baseline and at least one post-baseline assessment of the primary efficacy variable. Patients with a baseline x-ray and a 12M x-ray are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of participants | 0.9 | 2.8

3. Secondary Outcome: Percentage of Participants With at Least One New Moderate or Severe Morphometric Vertebral Fracture Over 12 Months
Description: Moderate or severe vertebral fracture (VF) was assessed based on morphometry. A QM (quantitative morphometry) incident VF(QM positive) was defined by at least a 20% decrease in any vertebral height (at least 4 mm). If a participant had a QM positive at any vertebrae at any visit,x-rays from all visits for participants were evaluated using Genant semi-quantitative (SQ) method for VF assessment. Grade 2 moderate VF was defined as a 25-40% reduction in any vertebral height.Grade 3 Severe: VF was defined as more than 40% reduction in any vertebral height.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of participants | 0.4 | 1.9

4. Secondary Outcome: Percentage of Participants With at Least One New Moderate or Severe Morphometric Vertebral Fracture Over 24 Months
Description: as for outcome 3
Time Frame: 24 Months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of participants | 1.1 | 3.0

5. Secondary Outcome: Percentage of Participants With at Least One New or Worsening Morphometric Vertebral Fracture Over 12 Months
Description: Worsening vertebral fracture (VF) was assessed based on morphometry. QM (quantitative morphometry) incident VF(QM positive) was defined by at least a 20% decrease in any vertebral height (at least 4 mm). If a participant had a QM positive at any vertebrae at any visit, x-rays from all visits for participants were evaluated using Genant semi-quantitative (SQ) method for VF assessment. A worsening fracture was defined as an SQ reading that was greater than the baseline SQ reading, which was at least 1 (prevalent fracture)
Time Frame: Baseline, 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of Participants | 1.3 | 2.8

6. Secondary Outcome: Percentage of Participants With at Least One New or Worsening Morphometric Vertebral Fracture Over 24 Months
Description: Worsening vertebral fracture (VF) was assessed based on morphometry. A QM (quantitative morphometry) incident VF(QM positive) was defined by at least a 20% decrease in any vertebral height (at least 4 mm). If a participant had a QM positive at any vertebrae at any visit,x-rays from all visits for participants were evaluated using Genant semi-quantitative (SQ) method for VF assessment. A worsening fracture was defined as an SQ reading that was greater than the baseline SQ reading, which was at least 1 (prevalent fracture)
Time Frame: Baseline, Month 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 553 | 574
Percentage of Participants | 2.0 | 4.9

7. Secondary Outcome: Mean Change in Height From Baseline
Description: Height was measured using a stadiometer. Two measurements were taken in millimeters (mm), and repeated if the two measurements differed by greater than 4 mm. The average of the two (or four) height measurements was used for analysis
Time Frame: from Baseline to 12 months and 24 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mm
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 529 | 547
mm
  12 months | -0.86 (0.333) | -2.50 (0.522)
  24 months | -2.33 (0.389) | -4.61 (0.610)

8. Secondary Outcome: Number of Participants With First Clinical Vertebral Fracture
Description: Clinical vertebral fracture is a painful vertebral fracture which came to clinical attention, e.g., with increased back pain, impairment of mobility or functional limitations. Subjects who did not experience a fracture event were censored at the end of study. End of study was defined as the last visit or date of death, whichever was earlier.
Time Frame: 24 months
Population: The ITT (intent to treat) population consisted of all subjects as randomized.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 588 | 611
Participants | 1 (NA) | 3 (1.63)

9. Secondary Outcome: Number of Participants With First Clinical Fracture
Description: Clinical fracture is painful fracture in any site which came to clinical attention, e.g., with increased pain, impaired mobility or functional limitations. Subjects who did not experience fracture were censored at end of study. End of study was defined as the earlier of last visit or date of death.
Time Frame: 24 months
Population: The ITT (intent to treat) population consisted of all subjects as randomized.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 588 | 611
Participants | 6 (1.95) | 11 (3.09)

10. Secondary Outcome: Number of Participants With First Non-vertebral Fracture
Description: Non-vertebral fracture is any fracture which was not of the vertebrae. Subjects who did not experience a fracture event were censored at the end of study. End of study was defined as the last visit or date of death, whichever was earlier.
Time Frame: 24 months
Population: The ITT (intent to treat) population consisted of all subjects as randomized.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 588 | 611
Participants | 5 (1.88) | 8 (2.83)

11. Secondary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Mass Density (BMD)
Description: Dual energy x-ray absorptiometry (DXA) Least Square Means (LSM) were analyzed using an ANCOVA model with treatment and baseline value as explanatory variables. Percent change in BMD at lumbar spine at Months 6, 12, and 24 relative to baseline as measured by DXA in a subset of at least 100 evaluable subjects at selected sites. Percentage change from baseline = 100*(endpoint - baseline)
Time Frame: Month 6, Month 12, Month 24
Population: Intent-to-treat (ITT) population included all randomized subjects who had a baseline and at least one post-baseline assessment of the efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: Percent change in BMD
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 65 | 63
Percent change in BMD
  Month 6 (n=61, n=61) | 4.87 (0.412) | 0.10 (0.412)
  Month 12 (n=60, n=62) | 5.51 (0.437) | 0.84 (0.430)
  Month 24 (n=58, n=61) | 7.73 (0.459) | 1.61 (0.448)

12. Secondary Outcome: Percentage Change From Baseline in Total Hip BMD (g/CM^2)
Description: Dual energy x-ray absorptiometry (DXA) Least Square Means (LSM) were analyzed using an ANCOVA model with treatment and baseline value as explanatory variables. Percent change in total hip BMD at Months 6, 12, and 24 relative to baseline as measured by DXA in a subset of at least 100 evaluable subjects at selected sites. Percentage change from baseline = 100*(endpoint - baseline)
Time Frame: Month 6, Month 12, Month 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percent change in BMD
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 64 | 65
Percent change in BMD
  Month 6 (n=60, n=63) | 1.38 (0.294) | -0.44 (0.287)
  Month 12 (n=58, n=64) | 1.66 (0.283) | 0.26 (0.269)
  Month 24 (n=56, n=63) | 2.31 (0.346) | 0.16 (0.326)

13. Secondary Outcome: Percentage Change From Baseline in Femoral Neck BMD (g/CM^2)
Description: Dual energy x-ray absorptiometry (DXA) Least Square Means (LSM) were analyzed using an ANCOVA model with treatment and baseline value as explanatory variables. Percent change in total femoral neck BMD at Months 6, 12, and 24 relative to baseline as measured by DXA in a subset of at least 100 evaluable subjects at selected sites. Percentage change from baseline = 100*(endpoint - baseline)
Time Frame: Month 6, Month 12, Month 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percent change in BMD
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 64 | 65
Percent change in BMD
  Month 6 (n=60, n=63) | 2.21 (0.448) | 0.58 (0.437)
  Month 12 (n=58, n=64) | 2.06 (0.465) | 0.59 (0.443)
  Month 24 (n=56, n=63) | 3.39 (0.544) | 0.09 (0.513)

14. Secondary Outcome: Serum Beta C-terminal Telopeptides of Type I Collagen(b-CTx) by Visits
Time Frame: Baseline, Month 3, Month 6, Month 12, Month 15, month 18, Month 24
Population: The ITT, Intent to Treat population, includes all participants who received a single a dose of treatment and had data available for analysis. n = the number of subjects with evaluable measurements at visit, as determined by the efficacy window.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 64 | 66
ng/mL
  Baseline (n-64) (n=66) | 0.3646 (0.02094) | 0.3933 (0.02955)
  Month 3 (n=63) (n=65) | 0.0990 (0.00800) [0.22 to 0.31] | 0.3647 (0.02989) [0.22 to 0.31]
  Month 6 (n=62) (n=64) | 0.1384 (0.00914) [0.34 to 0.47] | 0.3540 (0.02576) [0.34 to 0.47]
  Month 12 (n=63) (n=64) | 0.1669 (0.00925) [0.38 to 0.53] | 0.4042 (0.03056) [0.38 to 0.53]
  Month 15 (n=55) (n=58) | 0.0996 (0.00590) | 0.3576 (0.02519)
  Month 18 (n=55) (n=60) | 0.1320 (0.00661) | 0.3954 (0.03001)
  Month 24 (n=55) (n=62) | 0.1760 (0.01248) [0.38 to 0.52] | 0.4060 (0.02640) [0.38 to 0.52]

ADVERSE EVENTS:
Groups:
- Zoledronic Acid: 5 mg/100 ml administered via a peripheral intravenous site as a slow infusion over 15 minutes. The i.v. infusion was delivered via vented infusion line (to allow constant flow) and 20-22 gauge angiocatheter, and preceded and followed by a 10 ml normal saline flush of the intravenous line for a total volume infused of 120 ml once a year
Arm/Group | Zoledronic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 149/588 | 154/611
Other Adverse Events (participants affected / at risk) | 399/588 | 256/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=588) | Placebo (N=611)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 1
Angina pectoris (Cardiac disorders) | 6 | 7
Angina unstable (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 5
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 4
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Exomphalos (Congenital, familial and genetic disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Heterophoria (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal congestion (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 2
Death (General disorders) | 1 | 2
Device failure (General disorders) | 1 | 0
Device occlusion (General disorders) | 0 | 2
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 4
Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 9
Pyelonephritis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 16 | 10
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 4 | 5
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcohol induced persisting dementia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Brain compression (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 5
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cervical root pain (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 4 | 3
Depression (Psychiatric disorders) | 1 | 0
Encopresis (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urethral polyp (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Walking disability (Social circumstances) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 1
Arteritis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 1
Intermittent claudication (Vascular disorders) | 1 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 2
Varicose vein (Vascular disorders) | 0 | 1
Vascular calcification (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=588) | Placebo (N=611)
Chills (General disorders) | 40 | 5
Fatigue (General disorders) | 40 | 13
Influenza like illness (General disorders) | 30 | 14
Pyrexia (General disorders) | 143 | 21
Influenza (Infections and infestations) | 30 | 28
Nasopharyngitis (Infections and infestations) | 50 | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 123 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 82 | 73
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 30 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 129 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 23
Headache (Nervous system disorders) | 80 | 27
Hypertension (Vascular disorders) | 47 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.